CLINICAL TRIAL: NCT03680703
Title: Randomized Clinical Trial Testing Two Scalable Internet-Based Weight Loss Treatments Following Bariatric Surgery
Brief Title: Bariatric Scalable Internet Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000023155
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Bariatric Surgery; Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet (Experimental): Guided self-help behavioral weight loss treatment delivered via the internet
  Interventions: Behavioral: Guided Self-Help Behavioral Weight Loss
- Internet Plus Phone (Experimental): Guided self-help behavioral weight loss treatment delivered via the internet with weekly phone consultations
  Interventions: Behavioral: Guided Self-Help Behavioral Weight Loss

INTERVENTIONS:
Behavioral: Guided Self-Help Behavioral Weight Loss — Participants will be provided with patient-focused materials and worksheets that contain all the necessary information, procedures, and techniques of the behavioral weight loss program. For 12 weeks, treatment will be provided over the internet. This therapy focuses on making gradual and modest lifestyle changes with goals of normalizing eating patterns, decreasing caloric intake, building coping skills, and increasing physical activity.

SUMMARY:
The purpose of the study is to conduct a randomized clinical trial examining the feasibility and effectiveness of two guided self-help behavioral weight loss (gshBWL) treatments delivered via the internet for individuals struggling with weight loss one year following bariatric surgery. The two treatments will consist of 1) gshBWL delivered through the internet only (gshBWL-I) and 2) gshBWL delivered via the internet with additional complementary phone sessions (gshBWL-IP).

ELIGIBILITY:
Inclusion Criteria:

* gastric bypass and sleeve surgery patients from Yale's Bariatric/Gastrointestinal Surgery Program
* surgery 1-2 years prior
* <60% excess weight loss
* able to read English proficiently enough to read the patient self-help materials and study assessments
* available for the duration of the treatment
* availability of internet and phone to participate in study interventions
* agree to the study procedures

Exclusion Criteria:

* medical status judged by the surgeon as contraindication (rare instances of need for additional surgery or medical instability)
* unable to ambulate
* current medications that influence eating/weight
* current substance dependence or other severe psychiatric disturbance (e.g., suicidality) that requires immediate treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Weight Change | 3 months
  Percent weight loss (in pounds) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Ivezaj, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Department of Psychiatry, New Haven, Connecticut, United States